CLINICAL TRIAL: NCT05472480
Title: Association Between Anthropometric and Psychosocial Measurements in Vascular Disease
Brief Title: Anthropometric and Psychosocial Measurements in Vascular Disease
Acronym: ANPSYSOMEVAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Catanzaro (Other)
Responsible Party: Principal Investigator, Prof. Raffaele Serra, MD, Ph.D., Associate Professor of Vascular Surgery, University of Catanzaro
Other Study IDs: E.R.ALL.2018.51
Record Dates: First submitted 2022-07-20; First posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Vascular Diseases; Psychosocial Problem; Social Functioning
Keywords: sociology; vascular disease; anthropometric measurements; Psychosocial
MeSH Terms: conditions — Vascular Diseases; Social Adjustment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Chronic Venous Disease Patients: Consecutive patients admitted to Vascular Surgery Units.
  Interventions: Diagnostic Test: anthropometric and psychosocial measurements
- Carotid Stenosis Patients: Consecutive patients admitted to Vascular Surgery Units.
  Interventions: Diagnostic Test: anthropometric and psychosocial measurements
- Abdominal Aortic Aneurysm Patients: Consecutive patients admitted to Vascular Surgery Units.
  Interventions: Diagnostic Test: anthropometric and psychosocial measurements
- Peripheral Artery Disease Patients: Consecutive patients admitted to Vascular Surgery Units.
  Interventions: Diagnostic Test: anthropometric and psychosocial measurements

INTERVENTIONS:
Diagnostic Test: anthropometric and psychosocial measurements — Different types of measurements will be evaluated: body mass index (BMI), weight, height, waist circumference, waist / hip ratio (WHR), waist / stature (WSR) and the ABSI "a body" score shape index ". To complete the study, the personal experiences of the patients will be analyzed through the administration of a psycho-social questionnaire, Body Image Disturbance Questionnaire (BIDQ).

SUMMARY:
This experimental study is to verify a possible correlation between vascular disease, and anthropometric, and psychosocial measurements.

Consecutive patients with vascular diseases (Chronic Venous Disease, Carotid Stenosis, Abdominal Aortic Aneurysm, Peripheral Artery Disease) will be referred to Vascular Surgery Units of two hospitals linked to Interuniversity Center of Phlebolymphology (CIFL) International Research and Educational Program in Clinical and Experimental Biotechnology (Mater Domini University Hospital of Catanzaro and the Federico II University Hospital of Naples) to be evaluated.

Since it is necessary to study the anthropometric measures and the psychosocial aspects, different types of measurements will be carried out in order to correlate them with the aforementioned vascular disease.

DETAILED DESCRIPTION:
This is a cross sectional study with the aim analyze the association between the anthropometric and psychosocial measures in the following vascular disease: Chronic Venous Disease (CVD), Carotid Stenosis (CS) , Abdominal Aortic Aneurysm (AAA) , Peripheral Artery Disease (PAD).

Consecutive patients with vascular diseases (CVD, CS, AAA, PAD) referred to Vascular Surgery Units of two hospitals (Mater Domini University Hospital of Catanzaro and the Federico II University Hospital of Naples) will be evaluated.

Different types of measurements will be evaluated: body mass index (BMI), weight, height, waist circumference, waist / hip ratio (WHR), waist / stature (WSR) and the ABSI "a body" score shape index ". To complete the study, the personal experiences of the patients will be analyzed through the administration of a psycho-social questionnaire, Body Image Disturbance Questionnaire (BIDQ).

The data will be extrapolated from a prospective analysis on patients, by inserting in a Microsoft Excel database: demographic characteristics (age, sex); anthropometric parameters (height, weight, BMI, waist circumference WHR WSR ABSI); comorbidities, with particular reference to Diabetes mellitus, Dyslipidemia, Hypertension, CRI, coronary heart disease; smoking as a risk factor; the questionnaire for psychosocial aspects (BIDQ) on cumulative score (1-15); the vascular disease under examination. Population variables (age) and continuous outcomes (weight, age, BMI, waist circumference, WHR, WSR, ABSI, BIDQ) will be analyzed by Kruskal-Wallis test, while categorical variables (males, smokers, hypertension, diabetes, insulin-dependent diabetes, dyslipidemia, CAD, renal insufficiency) with Pearson's Chi-square test. The statistically significant outcomes will be subjected to sub-analysis with t-test, to identify the comparisons responsible for statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years, both genders, being a patient with one type of vascular disease at the time of the study.

Exclusion Criteria:

* presence of more than one contemporary vascular disease at the time of the study, to avoid overlapping of concomitant vascular disease.
* presence of any illiteracy, or psychiatric issues that may impair understanding or self-administration of the questionnaire.
* malignancies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with vascular diseases (CVD, CS, AAA, PAD) admitted to Vascular Surgery Units of two hospitals linked with Interuniversity Center of Phlebolymphology (CIFL) International Research and Educational Program in Clinical and Experimental Biotechnology (Mater Domini University Hospital of Catanzaro and the Federico II University Hospital of Naples).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Analysis of BMI | 32 months
  This measurement (reported in kg/m^2) will be related to the presence of vascular disease
Analysis of waist circumference | 32 months
  This measurement (reported in cm) will be related to the presence of vascular disease
Analysis of waist / hip ratio (WHR) | 32 months
  This ratio will be related to the presence of vascular disease
Analysis of waist / stature (WSR) | 32 months
  This ratio will be related to the presence of vascular disease
Analysis of ABSI "a body" score shape index | 32 months
  This index (range: from "Less than -0.868" to "Greater than +0.798") will be related to the presence of vascular disease
Administration of a psycho-social questionnaire, Body Image Disturbance Questionnaire (BIDQ). | 32 months
  The BIDQ comprises seven items. Items 1-2 assess appearance concern and preoccupation, while item 3 measures perceived distress, and items 4-7 investigate functional impairment and avoidance

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Serra, M.D., Ph.D., Study Chair — University Magna Graecia of Catanzaro
Locations (1):
- University Magna Graecia of Catanzaro, Catanzaro, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhu Q, Wang XB, Yao Y, Ning CX, Chen XP, Luan FX, Zhao YL. Association between anthropometric measures and cardiovascular disease (CVD) risk factors in Hainan centenarians: investigation based on the Centenarian's health study. BMC Cardiovasc Disord. 2018 May 2;18(1):73. doi: 10.1186/s12872-018-0810-8. PMID 29716519
- [Background] Dhana K, Ikram MA, Hofman A, Franco OH, Kavousi M. Anthropometric measures in cardiovascular disease prediction: comparison of laboratory-based versus non-laboratory-based model. Heart. 2015 Mar;101(5):377-83. doi: 10.1136/heartjnl-2014-306704. Epub 2014 Dec 11. PMID 25502814
- [Background] Venkatrao M, Nagarathna R, Patil SS, Singh A, Rajesh SK, Nagendra H. A composite of BMI and waist circumference may be a better obesity metric in Indians with high risk for type 2 diabetes: An analysis of NMB-2017, a nationwide cross-sectional study. Diabetes Res Clin Pract. 2020 Mar;161:108037. doi: 10.1016/j.diabres.2020.108037. Epub 2020 Jan 29. PMID 32004696